CLINICAL TRIAL: NCT06416176
Title: The Effect of a Mindfulness-Based Stress Reduction Program On Fatigue, Self-Efficacy And Stress in Patients With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: The Effect of a Mindfulness-Based Stress Reduction Program in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acetinkaya002
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Mindfulness; Upper Motor Neuron Lesion
Keywords: Mindfulness; Multiple sclerosis; Fatigue; Self-efficacy
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group received an 8-week MBSR program by an MBSR instructor.
  Interventions: Other: Mindfulness-Based Stress Reduction (MBSR) Program
- Control group (No Intervention): The patients in the control group continued to visit the society for their scheduled examinations and controls; no intervention was given to them. Furthermore, the control group received an invitation to participate in an identical MBSR program session following the study's conclusion.

INTERVENTIONS:
Other: Mindfulness-Based Stress Reduction (MBSR) Program — Participants in the experimental group received an 8-week MBSR program by an MBSR instructor. Each meeting were planned as a 3-hour session that completes the mindfulness training procedures by doing an opening meditation of 30- 45 minutes about that week, after the information about the meeting topic of the week is discussed. Experiences after meditation were shared with the group. Each week, the meeting topic and meditation continued with different contents, and practice meditations on the subject were held every week and home exercises were given. Home practice meditations were performed by listening to the guide audio recording with headphones. All home exercises in the training content were followed up on a daily basis and recorded.
  Arms: Experimental group

SUMMARY:
The aim of this study is to investigate the effect of an mindfulness-based stress reduction (MBSR) program designed in accordance with the literature and the basic principles of the program on fatigue, self-efficacy and stress for individuals with multiple sclerosis (MS).

Thirty members of the Multiple Sclerosis Society with multiple sclerosis were randomized as experimental and control groups. Participants in the experimental group received an 8-week MBSR program by an MBSR instructor. The patients in the control group continued to visit the society for their scheduled examinations and controls; no intervention was given to them. Outcome measurements consisted of Fatigue Impact Scale (FIS), Self-Efficacy Scale and Perceived Stress Scale.

DETAILED DESCRIPTION:
The use of mindfulness-based interventions to reduce fatigue in individuals with MS is supported by meta-analytic evidence. A systematic review concluded that mindfulness-based interventions effectively improves the quality of life in MS patients. To characterize the best formatting, mechanisms of action, and outcomes in MS patients with a wider range of social, educational, and clinical backgrounds, more research is necessary.

Participants in the experimental group received an 8-week MBSR program by an MBSR instructor. Each meeting were planned as a 3-hour session that completes the mindfulness training procedures by doing an opening meditation of 30- 45 minutes about that week, after the information about the meeting topic of the week is discussed. Experiences after meditation were shared with the group. Each week, the meeting topic and meditation continued with different contents, and practice meditations on the subject were held every week and home exercises were given. Home practice meditations were performed by listening to the guide audio recording with headphones. All home exercises in the training content were followed up on a daily basis and recorded.

The patients in the control group continued to visit the society for their scheduled examinations and controls; no intervention was given to them. Furthermore, the control group received an invitation to participate in an identical MBSR program session following the study's conclusion.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsing-remitting MS or progressive MS
* over 18 years of age,
* neurologist confirmed diagnosis of MS,
* a score of less than or equal to 7.0 on the Expanded Disability Status Scale (EDSS).

Exclusion Criteria:

* comorbidities with life-threatening physical or mental health (such as active psychosis, suicidal ideation, or terminal or life-threatening co-occurring medical diseases), or disorders that are predicted to severely restrict participation and adherence (e.g., dementia, pregnancy, ongoing substance abuse);
* individuals who are presently undergoing non-pharmacological psychological treatments or prior formal training in mindfulness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Fatigue Impact Scale | at baseline and at week 8
  It is a multidimensional fatigue scale that is frequently used in clinical and experimental investigations to assess the impact of fatigue on the body, mind, and social interactions.
Self-Efficacy Scale | at baseline and at week 8
  The scale, which does not belong to any subjective domain, measures the general perception of self-efficacy.
Perceived Stress Scale | at baseline and at week 8
  The scale was developed by Cohen et al in 1983 . Consisting of 14 items in total, Perceived Stress Scale is designed to measure how stressful a person's life is perceived by certain situations.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Çetinkaya, PhD, Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No